CLINICAL TRIAL: NCT02532816
Title: The Effect of Higher Nutrient-Dense Complementary Foods on Catch-up Growth and Nutritional Status of Stunting Children in Dompu District, Indonesia
Brief Title: Nutrient-Dense Complementary Foods on Catch-up Growth and Nutritional Status of Stunting Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SEAMEO Regional Centre for Food and Nutrition (Other)
Collaborators: Nestlé Foundation (Other); Indonesia University (Other); Institut Pertanian Bogor (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Duma Octavia Fransisca, MSc, PhD candidate, SEAMEO Regional Centre for Food and Nutrition
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ind_dompustunting
Record Dates: First submitted 2015-08-20; First posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Stunting
Keywords: stunting; indonesia
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HND-CF (Experimental): subjects will receive nutrient dense complementary foods in optimized CFRs + fortified biscuit (ferrous fumarate 83.5 mg, zinc oxide 50.95 mg, Calcium carbonate 3104.05 mg, Thiamine Mononitrate1.85 mg, Nicotinic Acid 30.45 mg, Pyridoxine Hydrocloride 2.90 mg, Pteroyl monoglutamic acid 764.90 mcg, Cyanocobalamin 0.95 mcg, Retinol Palmitate (dry) 742.50 mcgRE)
  Interventions: Dietary Supplement: Nutrient dense complementary foods
- SND-CF (Active Comparator): subjects will receive nutrient dense complementary foods in optimized CFRs + fortified biscuit (ferrous fumarate 32.6 mg, zinc oxide 3.78 mg, Calcium carbonate 874.12 mg, Thiamine Mononitrate1.25 mg, Nicotinic Acid 17.95 mg, Pyridoxine Hydrocloride 1.10 mg, Pteroyl monoglutamic acid 329.90 mcg, Cyanocobalamin 0.55 mcg)
  Interventions: Dietary Supplement: Nutrient dense complementary foods
- NDN-CF (Placebo Comparator): subjects will receive nutrient dense complementary foods in optimized CFRs + non fortified biscuit
  Interventions: Dietary Supplement: Nutrient dense complementary foods

INTERVENTIONS:
Dietary Supplement: Nutrient dense complementary foods — Mothers/caregivers will receive optimized CFRs to improve children diets and fortified biscuits (3 types of biscuit) for 6 days per week (in 12 months).
  Nutrition eduction for mothers/caregivers. Monthly body weight and length/height measurements

SUMMARY:
The purpose of this study is to determine and compare the effect of higher nutrient-dense complementary foods and standard nutrient dense complementary foods on the catch-up growth and nutritional status of stunting children aged 12-23 months old in Indonesia.

DETAILED DESCRIPTION:
This is an intervention, double blind study. Investigators want to study the effect of higher nutrient density complementary foods (which consists of optimizing children diet by practicing Optimized Complementary Feeding Recommendation/CFRs and consume special designed fortified biscuit) on catch-up growth and nutritional status of stunting children aged 12 - 23 mos old.

There are two phases in this study.

Phase I: Development of CFRs and fortified biscuit

1. Food consumption survey (n=100) to gather information on foods typically consumed by the stunting children, food patterns, serving sizes, food price.

Methods: 24-hr dietary recall, food weighed dietary records (WDR) and 5-days food tally for each child.

Data from food consumption survey will be use to develop optimized CFRs by using Linear Programming (LP) approach with software Optifood v 2.0.

Data from LP analysis such as nutrient gaps will be use to formulate fortified biscuit (3 type of nutrient dense). Biscuit ingredients will use local foods. Acceptability trials will be conducted to see the acceptance of the biscuit in the community settings (color, smell, taste and portion).

Phase II: Intervention Screening: Anthropometry measurements (body weight and length) to screen stunting and non stunting children; and child with hemoglobine level < 7 g/dL was referred to sub-district health center.

Baseline survey: anthropometry measurements (body weight and length), biochemical assessments (3 mL of blood obtain from the antecunital vein for serum zinc, ferritin, transferin receptor, CRP, AGP and RBP), dietary assessment (repeated 24-h recall), socio-demography, food security, health seeking practices questionnaires.

Intervention -- optimized CFRs + Biscuits (3 groups) Biscuits will be distributed for 6 days consumption per week (12 months). The waste of the biscuits will be weighted to get actual biscuit consumptions. Mothers/caregivers will be encouraged to practice CFRs to improve child's nutritional adequacy. Monthly body weight and length/height measurement. Nutrition education for mothers/caregivers by field staff.

Endline survey: anthropometry measurements (body weight and length), biochemical assessments (3 mL of blood obtain from the antecunital vein for serum zinc, ferritin, transferin receptor, CRP, AGP and RBP), dietary assessment (repeated 24-h recall)

ELIGIBILITY:
Inclusion Criteria:

* identified as stunting (having HAZ ≤ -2SD of the WHO Growth Standard 2006)
* no clinical evidence of any acute infectious disease or other diseases or morbidity condition that could interfere with the intake of study diets
* parents and children residence in the study area.
* parental concent obtained

Exclusion Criteria:

* presence of oedema, severe illness warranting hospitalization on the enrolment day such as persistent diarrhea and other disease which may influence feeding practices and nutrient absorption
* conncurrent participation in another clinical trial
* severe anemia with hemoglobine concentration < 7.0 g/dL

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 217 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
length gain | one year
  The increment of body length/height of the subjects, monthly measurement
linear growth rate | one year
  growth velocity = (x2-x1)/(t2-t1) where x2 and x1 are values of the measurement on two occacions t2 and t1. in mm/d

CONTACTS AND LOCATIONS:
Overall Officials: Duma O Fransisca, MSc, Principal Investigator — SEAMEO Regional Centre for Food and Nutrition; Umi Fahmida, Dr, Principal Investigator — SEAMEO Regional Centre for Food and Nutrition
Locations (1):
- in the community (Woja,Manggelewa, Kempo subdistrict), Dompu, West Nusa Tenggara, Indonesia

REFERENCES:
- [Background] Golden MH. Proposed recommended nutrient densities for moderately malnourished children. Food Nutr Bull. 2009 Sep;30(3 Suppl):S267-342. doi: 10.1177/15648265090303S302. PMID 19998863
- [Background] Ferguson EL, Darmon N, Briend A, Premachandra IM. Food-based dietary guidelines can be developed and tested using linear programming analysis. J Nutr. 2004 Apr;134(4):951-7. doi: 10.1093/jn/134.4.951. PMID 15051853